CLINICAL TRIAL: NCT05521750
Title: Learning Curve, Outcome Parameters, and MRI Assessment Of Disc Evacuation After Transforaminal Percutaneous Endoscopic Lumbar Discectomy: a Single Center Retrospective Cohort Study
Brief Title: Learning Curve, Outcome Parameters, and MRI Assessment of Disc Evacuation After Transforaminal Percutaneous Endoscopic Lumbar Discectomy
Status: Completed | Type: Observational
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Yudha Mathan Sakti, Head of Orthopedic residency program, Gadjah Mada University, Yogyakarta, Indonesia, Gadjah Mada University
Other Study IDs: UGM_PELD
Record Dates: First submitted 2022-08-19; First posted 2022-08-30 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Herniated Nucleus Pulposus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Weight of Intervertebral disc which taken during TPELD in our institution hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (13):
- Age: Patient age
  Interventions: Procedure: Transforaminal Percutaneous Endoscopic Lumbar Decompression
- Gender: Patient's gender
  Interventions: Procedure: Transforaminal Percutaneous Endoscopic Lumbar Decompression
- Surgical Time: Duration of surgery, begin from incision until skin closure
  Interventions: Procedure: Transforaminal Percutaneous Endoscopic Lumbar Decompression
- Intraoperative Blood loss: Total blood loss during operation
  Interventions: Procedure: Transforaminal Percutaneous Endoscopic Lumbar Decompression
- Length of Stay: Duration of hospitalization
  Interventions: Procedure: Transforaminal Percutaneous Endoscopic Lumbar Decompression
- VAS Pre-op: Pain scale measured with visual analog scale (VAS) prior to the operation
  Interventions: Procedure: Transforaminal Percutaneous Endoscopic Lumbar Decompression
- 1 Month VAS: Pain scale measured with visual analog scale (VAS) 1 month after the operation
  Interventions: Procedure: Transforaminal Percutaneous Endoscopic Lumbar Decompression
- 3 Month VAS: Pain scale measured with visual analog scale (VAS) 3 month after the operation
  Interventions: Procedure: Transforaminal Percutaneous Endoscopic Lumbar Decompression
- Decrease VAS 1 month: Difference of VAS score within 1 month of evaluation
  Interventions: Procedure: Transforaminal Percutaneous Endoscopic Lumbar Decompression
- Decrease VAS 3 month: Difference of VAS score within 3 month of evaluation
  Interventions: Procedure: Transforaminal Percutaneous Endoscopic Lumbar Decompression
- Disc weight: Estimation of total disc weight
  Interventions: Procedure: Transforaminal Percutaneous Endoscopic Lumbar Decompression
- Removed disc weight: weight of removed disc measured after operation
  Interventions: Procedure: Transforaminal Percutaneous Endoscopic Lumbar Decompression
- Percentage of Removed Disc: Percentage of removed disc as seen on the axial MRI
  Interventions: Procedure: Transforaminal Percutaneous Endoscopic Lumbar Decompression

INTERVENTIONS:
Procedure: Transforaminal Percutaneous Endoscopic Lumbar Decompression — TPELD is procedure of percutaneous lumbar discectomy done under endoscopic setting
  Other Names: TPELD

SUMMARY:
Transforaminal Percutaneous Endoscopic Lumbar Discectomy (TPELD) is a surgical technique for managing lumbar disc herniation. The procedure demands a steep learning curve with regards to clinical improvement and technical challenges for disc evacuation. This study was to evaluate learning curve, outcome parameters, and MRI assessment for successful procedure in single - center early experience of Transforaminal Percutaneous Endoscopic Lumbar Discectomy (TPELD).

This study was a retrospective cohort study, involving patients who underwent TPELD in our institution hospital by a single surgeon.

DETAILED DESCRIPTION:
Investigators reviewed clinical evaluation, C-arm shot, and post-operative MRI findings as parameters for evaluation. All data was taken from the patients' medical records with single-level LDH (Lumbar Disc Herniation) following TPELD. Patients with incomplete data and those who underwent revision surgery were excluded. The collected data were regarding the sociodemographic characteristics of the patients (age and gender), surgical time, pre-operative pain scale (1-10), postoperative pain scale, complications, and weight of the removed disc and ODI (Oswestry Disability Index) score. The preoperative pain scale was assessed within 48 hours before the surgery while the post-operative pain scale was assessed at one month and three months after the surgery. The reduction of pain was assessed, comparing the pre-operative pain scale and the post-operative pain scale at 1 month and 3 months follow up.

Pre TPELD MRI data and 3 months post TPELD were collected to evaluate the percentage of disc removed referring to the quantification of the axial MRI by two independent radiology department personnel. The area of the bulging disc was measured using as many points as the user felt were necessary in order to trace a reasonable outline of disc herniation.

All of the TPELD procedures are performed by a single spine surgeon with only using one type of endoscopic instrumentation in one level LDH. The surgeon was not involved during data collection and data were collected by independent assessors.

The statistical analysis was performed using SPSS 23.0. investigator tested all the numeric variables with the Shapiro-Wilk test for the normality of distribution. The surgeon's learning curve was evaluated using negative curve-fit regression analysis (y = ae-bx+ c) described by Silva, et al (2013). Then all case are divided into two groups based on the surgical time: cases before and at reaching 50% proficiency (early group) and cases after reaching 50% proficiency (later group).

ELIGIBILITY:
Inclusion Criteria:

* patient with single level LDH
* treated with TPELD

Exclusion Criteria:

* reoperation
* inclomplete medical record

Ages: 24 Years to 62 Years | Sex: All
Age Groups: Adult
Study Population: Patient with LDH under orthopedic spine division of RSUP dr. Sarjito Jogjakarta
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2021-06-06 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Learning curve of surgeon based on the duration | measured within 24 hours after procedure is done
  Curve of milestone achieved by the surgeon in performing the procedyre
Learning curve based on removed disc | measured within 24 hours after procedure is done
  Curve of milestone achieved by the surgeon based on extracting targeted disc weight
Learning curve based on the C-arm shot | measured within 24 hours after procedure is done
  Curve of milestone achieved by the surgeon based on use of fluoroscopic imaging

SECONDARY OUTCOMES:
Pain reduction after one month | 1 month after procedure
  We measured the pain with visual analog score (VAS) scale reduction on each patients (1-10)
Pain reduction after three month | 3 month after procedure
  We measured the pain with visual analog score (VAS) scale reduction on each patients (1-10)

CONTACTS AND LOCATIONS:
Locations (1):
- RSUP dr. Sarjito, Sleman, DIY, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided